CLINICAL TRIAL: NCT03495635
Title: Randomized Controlled Trial of the Big Brothers Big Sisters Community-Based Mentoring Program for Prevention of Crime and Juvenile Delinquency
Brief Title: Randomized Controlled Trial of Big Brothers Big Sisters Mentoring for Prevention of Crime and Delinquency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Laura and John Arnold Foundation (Other); Herrera Consulting Group, LLC (Unknown); Big Brothers Big Sisters of America (Unknown); National Council of Juvenile and Family Court Judges (Unknown)
Responsible Party: Principal Investigator, David DuBois, Professor of Community Health Sciences, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017-0291
Record Dates: First submitted 2018-01-04; First posted 2018-04-12 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Crime; Juvenile Delinquency
Keywords: mentoring; prevention

STUDY DESIGN:
Intervention Model Description: Enrolled participants will be assigned randomly to participate in the Big Brothers Big Sisters Community-Based Mentoring Program (treatment group) or to a wait-list control group that is not eligible to participate in the program for a period of 4 years.
Who Masked: Investigator
Masking Description: The research team will collect the 18-month follow-up surveys from participating youth and parents; masking of study condition will not be feasible for data collection staff, but primary study analyses will be conducted by the investigators with study condition masked. Juvenile justice authorities providing arrest record information will be masked to study arm of participants as will all those on the research team who are involved in coding this information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BBBS Community-Based Mentoring (Experimental): Big Brothers Big Sisters Community-Based Mentoring Program
  Interventions: Behavioral: Big Brothers Big Sisters Community-Based Mentoring Program
- Control (No Intervention): Not eligible to participate in a Big Brothers Big Sisters mentoring program, but may participate in other mentoring programs.

INTERVENTIONS:
Behavioral: Big Brothers Big Sisters Community-Based Mentoring Program — One-to-one mentoring provided by an adult volunteer with training and ongoing monitoring and support from program staff.
  Arms: BBBS Community-Based Mentoring

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the Big Brothers Big Sisters of America (BBBSA) community-based mentoring (CBM) program for prevention of crime and delinquency/conduct problems, including risk and protective factors for these outcomes. Approximately 2,500 youth ages 10-16 will be randomly assigned to either the CBM program or an untreated control group. Study outcomes will be assessed over a 4-year period via both youth- and parent-report surveys and official records of police/court contact (e.g., arrests).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of the Big Brothers Big Sisters of America (BBBSA) community-based mentoring (CBM) program for prevention of crime and delinquency/conduct problems, including risk and protective factors for these outcomes. Participants will be recruited from 16 BBBSA affiliates, which are located in different regions of the U.S. and were invited to serve as sites for the study using a random selection process. The study sample will consist of approximately 2,500 youth ages 10-16 whose parents seek services from one of the participating BBBSA affiliates during the study enrollment period and for whom consent/assent to participate in the research is obtained. Enrolled youth will be randomly assigned to participate in the CBM program (treatment group) or to a control group (no BBBSA programming during the youth's 4-year period of study participation). Youth will be assigned in a 3:1 ratio to the treatment and control groups. Youth and parents will complete survey measures both at study enrollment, prior to notification of assignment to control or treatment group, and 18 months later. Official records of police/court contact (e.g., arrests), with separate parent/guardian consent as provided at study enrollment, will be obtained both for the period preceding each youth's enrollment in the study and for a 4-year period following enrollment.

The study has 4 specific aims:

1. To determine the effects of participation in the Big Brothers Big Sisters CBM program on youth offending as measured by police/court records, i.e., person offense, property offense, drug law violation, public order offense, or status offense.
2. To determine the effects of participation in the BBBS CBM program on the likelihood of youths' involvement in delinquent behavior/conduct problems as assessed by youth and parent reports.
3. To determine the effects of BBBS CBM program participation on the likelihood of youths' involvement in substance use as assessed by self-reports of alcohol use to point of drunkenness, tobacco, or illicit drug use.
4. To determine the effects of BBBS CBM program participation on both risk and protective factors for delinquent/criminal behavior, such as aggression, depressive symptoms, association with deviant peers, self-control, and school connectedness, as assessed by youth and/or parent reports, and to explore the role of these effects in mediating effects of program participation on offending, delinquent behavior, and substance use.

ELIGIBILITY:
Inclusion criteria:

* youth is 10 years of age or older
* youth is likely to be eligible for the Big Brothers Big Sisters Community-Based Mentoring program as determined by initial assessment of program staff

Exclusion criteria:

* youth has a severe learning, cognitive or other intellectual disability as reported by the parent
* parent does not both speak and read either English or Spanish
* youth does not have a sibling who is already a study participant
* youth has been matched with a Big Brother/Sister through one of the affiliate's programs in the past
* youth has a sibling currently receiving services from the affiliate for whom services were initiated (i.e., inquiry was made) prior to start of the study
* youth belongs to a group that the affiliate is excluding from study participation based on previous agreement with the research team
* youth is designated as an exception case by affiliate staff (each affiliate will have the opportunity to exclude up to 4% of study-eligible youth from the research prior to consent and random assignment for any reason deemed appropriate (e.g., perceived high need of the youth))

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1361 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Arrest | 4 years
  0/1 indicator based on official police/court/juvenile office records of any of the following types of offenses-person offense, property offense, drug law violation, public order offense, or status offense
Arrest | 18 months
  0/1 indicator based on official police/court/juvenile office records of any of the following types of offenses-person offense, property offense, drug law violation, public order offense, or status offense
Delinquency | 18 months
  0/1 indicator based on youth and parent report using 13 items from the Add Health Study (Bearman et al., 1997)
Substance use | 18 months
  0/1 indicator based on youth report of alcohol use to point of drunkenness, tobacco, or illicit drug use

SECONDARY OUTCOMES:
Truancy | 18 months
  3-item youth-report measure (2 items from Herrera et al., 2013)
Association with deviant peers | 18 months
  A single measure computed as the average of scores on continuous youth-report measure (Elliott et al., 1996) and one-item (0/1) parent-report indicator from Youth Risk Index (Herrera et al., 2013) after each score has been standardized to mean of 0 and standard deviation of 1.
School suspensions | 18 months
  One-item (0/1) parent-report indicator from Youth Risk Index (Herrera et al., 2013)
Depressive symptoms | 18 months
  Depressive Symptoms Pediatric Self-Report - Short Form from the Patient-Reported Outcomes Measurement Information System (PROMIS) (Irwin et al., 2010). Lower scores indicate a better outcome
Impulsivity | 18 months
  A single measure computed as the average of scores on continuous youth- and parent-report scales (Hay & Meldrum, 2010) after each score has been standardized to mean of 0 and standard deviation of 1.
Conventional values | 18 months
  Belief in the Moral Order scale of the Communities That Care Youth Survey (Arthur et al., 2002)
Aggressive behavior | 18 months
  A single measure computed as the average of scores on youth-report Aggression Scale (Orpinas & Frankowski, 2001) and parent-report Parent's Checklist from the Fast Track Project: https://fasttrackproject.org/techrept/p/pcl/ after each score has been standardized to mean of 0 and standard deviation of 1.
Academic success | 18 months
  4-item measure of grades in core subjects (Herrera et al., 2013)
Positive parenting | 18 months
  Parent-report Positive Parenting subscale from the Alabama Parenting Questionnaire (Essau et al., 2006)
Parent involvement | 18 months
  Parent-report Involvement subscale from the Alabama Parenting Questionnaire (Essau et al., 2006)
Parental monitoring and supervision | 18 months
  Parent-report Poor Monitoring/Supervision subscale from the Alabama Parenting Questionnaire (Essau et al., 2006)
Parental consistent discipline | 18 months
  Parent-report Inconsistent Discipline subscale from the Alabama Parenting Questionnaire (Essau et al., 2006)
Family relationships | 18 months
  Parent-report General Functioning scale of the Family Assessment Device (Epstein et al., 1983)
Perceived social support from family members | 18 months
  Youth-report Multidimensional Scale of Perceived Social Support (Zimet et al., 1988): Family Members subscale
Perceived social support from peers | 18 months
  Youth-report Multidimensional Scale of Perceived Social Support (Zimet et al., 1988): Peers subscale
Perceived social support from special person | 18 months
  Youth-report Multidimensional Scale of Perceived Social Support (Zimet et al., 1988): Significant Others subscale
School engagement | 18 months
  Youth-report Behavioral Engagement subscale of the Engagement versus Disaffection with Learning Scale (Skinner et al., 2009)
Goal-setting and pursuit | 18 months
  Parent-report Goal Orientation scale from Child Trends: https://www.childtrends.org/research/research-by-topic/positive-indicators-project/goal-orientation/
Involvement in out-of-school-time activities | 18 months
  Parent-report (Herrera et al., 2007)
Volunteering in the community | 18 months
  Youth-report single-item (Herrera et al., 2013)
Life satisfaction | 18 months
  Youth-report single-item measure from WHO's 2005-06 Health Behaviors in School Age Children Survey: http://filer.uib.no/psyfa/HEMIL-senteret/HBSC/2006_Mandatory_Questionnaire.pdf
Self-esteem | 18 months
  Youth-report Global Self-Esteem subscale of brief version of the Self-Esteem Questionnaire (DuBois et al., 1996; Silverthorn et al., 2017)
Happiness | 18 months
  Youth-report Positive Affect Pediatric Self-Report - Short Form from the Patient-Reported Outcomes Measurement Information System (PROMIS) (Forrest et al., 2017)
Grit | 18 months
  Youth-report Grit Scale for Children (Duckworth & Quinn, 2009)
Social competence | 18 months
  Social Competencies Scale of the Youth Outcome Measures Online Toolbox (Muris, 2001)
Special interest development | 18 months
  Youth-report (adapted from DuBois & Keller, 2017)
Hopeful future expectations | 18 months
  Youth-report abbreviated version of the Hopeful Future Expectations Scale (Bowers et al., 2012)
Career exploration | 18 months
  Youth-report 2 items (adapted from Herrera et al., 2011)
College exploration | 18 months
  Youth-report 1 item (adapted from Herrera et al., 2011)
Self-advocacy | 18 months
  Youth-report (Jarjoura et al., 2017)
Coping efficacy | 18 months
  Youth-report 1 item adapted from Coping Efficacy Scale (Sandler et al., 2000)

CONTACTS AND LOCATIONS:
Overall Officials: David L DuBois, PhD, Principal Investigator — University of Illinois at Chicago; Carla Herrera, PhD, Principal Investigator — Herrera Consulting Group, LLC
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
At the study's conclusion, all individual participant data will be de-identified and made publicly available on the Open Science Framework website along with survey instruments and any code used to clean and analyze the data.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available August 2024 and will be permanently available thereafter
Access Criteria: Requests to access the IPD will be made in writing to the Principal Investigator and approved so long as there is a valid scientific rationale and appropriate IRB approval. The mechanism for sharing the data, all of which will be de-identified, will be secure and encrypted FTP and subject to approval of the PI's institutional IRB. Supporting information (see above list) will be available on the Open Science Framework at the web address below.
URL: https://osf.io/8ukfv/

REFERENCES:
- [Background] Arthur MW, Hawkins JD, Pollard JA, Catalano RF, Baglioni AJ Jr. Measuring risk and protective factors for substance use, delinquency, and other adolescent problem behaviors. The Communities That Care Youth Survey. Eval Rev. 2002 Dec;26(6):575-601. doi: 10.1177/0193841X0202600601. PMID 12465571
- [Background] Resnick MD, Bearman PS, Blum RW, Bauman KE, Harris KM, Jones J, Tabor J, Beuhring T, Sieving RE, Shew M, Ireland M, Bearinger LH, Udry JR. Protecting adolescents from harm. Findings from the National Longitudinal Study on Adolescent Health. JAMA. 1997 Sep 10;278(10):823-32. doi: 10.1001/jama.278.10.823. PMID 9293990
- [Background] Bowers, E. P., Geldhof, G. J., Schmid, K. L., Napolitano, C. M., Minor, K., & Lerner, J. V. (2012). Relationships with important nonparental adults and positive youth development: An examination of youth self-regulatory strengths as mediators. Research in Human Development, 9, 298-316. http://dx.doi.org/10.1080/15427609.2012.729911
- [Background] DuBois, D. L., Felner, R. D., Brand, S., Phillips, R. S. C., & Lease, A. M. (1996). Early adolescent self-esteem: A developmental-ecological framework and assessment strategy. Journal of Research on Adolescence, 6, 543-579.
- [Background] DuBois DL, Keller TE. Investigation of the Integration of Supports for Youth Thriving Into a Community-Based Mentoring Program. Child Dev. 2017 Sep;88(5):1480-1491. doi: 10.1111/cdev.12887. Epub 2017 Jun 19. PMID 28626886
- [Background] Duckworth AL, Quinn PD. Development and validation of the short grit scale (grit-s). J Pers Assess. 2009 Mar;91(2):166-74. doi: 10.1080/00223890802634290. PMID 19205937
- [Background] Essau, C. A., Sasagawa, S., & Frick, P. J. (2006). Psychometric properties of the Alabama Parenting Questionnaire. Journal of Child and Family Studies, 15, 597-616.
- [Background] Epstein, N. B., Baldwin, L. M., & Bishop, D. S. (1983). The McMaster Family Assessment Device. Journal of Marital and Family Therapy, 9, 171-180.
- [Background] Herrera C, Grossman JB, Kauh TJ, McMaken J. Mentoring in schools: an impact study of big brothers big sisters school-based mentoring. Child Dev. 2011 Jan-Feb;82(1):346-61. doi: 10.1111/j.1467-8624.2010.01559.x. PMID 21291446
- [Background] Herrera, C., Linden, L. L., Arbreton, J. A. & Grossman, J. B. (2011). Testing the impact of Higher Achievement's year-round out-of-school-time program on academic outcomes. Philadelphia: Public/Private Ventures.
- [Background] Irwin DE, Stucky B, Langer MM, Thissen D, Dewitt EM, Lai JS, Varni JW, Yeatts K, DeWalt DA. An item response analysis of the pediatric PROMIS anxiety and depressive symptoms scales. Qual Life Res. 2010 May;19(4):595-607. doi: 10.1007/s11136-010-9619-3. Epub 2010 Mar 7. PMID 20213516
- [Background] Jarjoura, G. R. et al. (2017). The Evaluation of The Mentoring Enhancement Demonstration Program. Washington, DC: American Institutes for Research. Manuscript in preparation.
- [Background] Muris, P. (2001). A brief questionnaire for measuring self-efficacy in youths. Journal of Psychopathology and Behavioral Assessment, 23, 145-149. http://dx.doi.org/10.1023/A:1010961119608
- [Background] Orpinas P, & Frankowski R. (2001). The aggression scale: a self-report measure of aggressive behavior for young adolescents. Journal of Early Adolescence, 21, 51-68.
- [Background] Sandler IN, Tein JY, Mehta P, Wolchik S, Ayers T. Coping efficacy and psychological problems of children of divorce. Child Dev. 2000 Jul-Aug;71(4):1099-118. doi: 10.1111/1467-8624.00212. PMID 11016569
- [Background] Bavarian N, Lewis KM, Acock A, DuBois DL, Yan Z, Vuchinich S, Silverthorn N, Day J, Flay BR. Effects of a School-Based Social-Emotional and Character Development Program on Health Behaviors: A Matched-Pair, Cluster-Randomized Controlled Trial. J Prim Prev. 2016 Feb;37(1):87-105. doi: 10.1007/s10935-016-0417-8. PMID 26781590
- [Background] Skinner, E. A., Kindermann, T. A., & Furrer, C. J. (2009). A motivational perspective on engagement and disaffection: Conceptualization and assessment of children's behavioral and emotional participation in academic activities in the classroom. Educational and Psychological Measurement, 69, 493-525. http://dx.doi.org/10.1177/0013164408323233
- [Background] Zimet, G. D., Dahlem, N. W., Zimet, S. G., & Farley, G. K. (1988). The Multidimensional Scale of Perceived Social Support. Journal of Personality Assessment, 52, 30-41. http://dx.doi.org/10.1207/s15327752jpa5201_2
- [Background] Elliott, D. S., Wilson, W. J., Huizinga, D., Sampson, R. J., Elliott, A., & Rankin, B. (1996). The effects of neighborhood disadvantage on adolescent development. Journal of Research in Crime and Delinquency, 33, 389. doi:10.1177=0022427896033004002
- [Background] Forrest CB, Ravens-Sieberer U, Devine J, Becker BD, Teneralli R, Moon J, Carle A, Tucker CA, Bevans KB. Development and Evaluation of the PROMIS(R) Pediatric Positive Affect Item Bank, Child-Report and Parent-Proxy Editions. J Happiness Stud. 2018 Mar;19(3):699-718. doi: 10.1007/s10902-016-9843-9. Epub 2017 Jan 21. PMID 29760578
- Available data/document: Individual Participant Data Set: osf.io/8ukfv — https://osf.io/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/35/NCT03495635/Prot_SAP_000.pdf